CLINICAL TRIAL: NCT02408419
Title: Proximal Obturator Nerve Block After Insufficient Analgesic Effect of Femoral Nerve Block in Patients With Hip Fracture
Brief Title: Obturator Nerve Block in Patients With Hip Fracture
Acronym: OPAD
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was completely redesigned
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: protocol2tdn
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-03

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Local anesthetic (Experimental): 15 ml. of local anesthetic
  Interventions: Drug: Bupivacaine
- Saline (Placebo Comparator): 15 ml. of saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Bupivacaine — Bupivacaine is injected proximally to anesthetize the obturator nerve
  Arms: Local anesthetic
Drug: Saline — Saline is injected as a placebo
  Other Names: Solution of sodium chloride
  Arms: Saline

SUMMARY:
About 10-30% of all patients with hip fracture have only insufficient analgesic effect of a femoral nerve block. One of the possible causes of this failure to provide analgesia from a single nerve block could be the that other nerves occasionally are involved in transmitting the pain signal. One of the nerves that is believed to give off branches to the hip is the obturator nerve.

With ultrasound it is possible to make a selective proximal nerve block of the obturator nerve.

The aim of this trail is to give patients with hip fracture and only insufficient effect of a femoral nerve block a supplementary obturator nerve block in a randomized manner with either local anesthetics or placebo in order to access the preoperative analgesic effect.

DETAILED DESCRIPTION:
About 10-30% of all patients with hip fracture have only insufficient analgesic effect of a femoral nerve block. One of the possible causes of this failure to provide analgesia from a single nerve block could be the that other nerves occasionally are involved in transmitting the pain signal. One of the nerves that is believed to give off branches to the hip is the obturator nerve. Earlier it was believed that the so called '3-in-1-block' or the iliac fascia compartment block would anesthetize also the obturator nerve, and these two nerve blocks have been uses extensively in the emergency ward for preoperative analgesia. Today that is not believed to be true and consequently is the part of the obturator nerve in patients with hip fracture unknown.

With ultrasound it is possible to make a selective proximal nerve block of the obturator nerve before it branches into an anterior and a posterior branch. A selective nerve block af the obturator nerve to access its effect in patients with hip fracture has to our knowledge never been done.

The aim of this trail is to give patients with hip fracture and only insufficient effect of a femoral nerve block a supplementary obturator nerve block in a randomized manner with either local anesthetics or placebo in order to access the preoperative analgesic effect.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of hip fracture
* Successful sensory cutaneous effect of the femoral nerve block
* Age ≥ 55 years
* Mentally capable of comprehending and using verbal pain score
* Mentally capable of differentiating between pain from the fractured hip and pain from other locations
* Mentally capable of understanding the given information
* Arrival in the emergency room at times when one of the doctors who do the nerve blocks for this investigation are on call
* Possible sonographic visualization of the structures needed for the nerve block
* Verbal numeric pain scale score (NRS 0-10) > 5 with passive leg raise of the fractured leg at the time of inclusion OR NRS > 3 at rest, 30 minutes after a femoral nerve block
* Patients informed consent

Exclusion Criteria:

* Hip fracture not confirmed by x-ray
* Weight < 45 kg
* Patient has previously been included in this trial
* If the patient wishes to be excluded
* Allergy to local anesthetics or adrenocortical hormone
* Visible infection in the area of the point of needle injection

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Success rate of successful analgesia | 20 minutes
  Success rate of successful analgesia 20 minutes after a supplementary obturator nerve block in patients with hip fracture

SECONDARY OUTCOMES:
Time used for the procedure | Expected average of 5 minutes
  Time from start of ultrasound scanning to end of injection of local anesthetic or placebo
Success rate of possible sonographic visualization | Expected average of 5 minutes
  Success rate of possible sonographic visualization of necessary anatomical structures i order to do the nerve block
Time to analgesia | 20 minutes
  Time from end of injection of local anesthetic to analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F. Bendtsen, MD, Ph.d., Study Director — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Aarhus, Denmark

REFERENCES:
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043